CLINICAL TRIAL: NCT03178942
Title: A Randomized, Double-Blind, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Permethrin Cream, 5% (Encube Ethicals) Compared to Elimite™ Cream (Permethrin) 5% (Prestium Pharma, Inc.) in the Treatment of Scabies
Brief Title: Multiple-Site Study to Evaluate the Therapeutic Equivalence of Permethrin Cream, 5% in the Treatment of Scabies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Encube Ethicals Pvt. Ltd. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71675502
Record Dates: First submitted 2017-05-31; First posted 2017-06-07 (Actual); Results first posted 2019-03-14 (Actual); Last update posted 2019-03-26 (Actual); Status verified 2019-02

CONDITIONS: Scabies
MeSH Terms: conditions — Scabies | interventions — Permethrin

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to the test or reference permethrin to treat scabies.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study product will be randomized, packaged and blinded so that the packaging for both treatments look identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reference: Elimite™ Cream (Active Comparator): Reference: Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.)
  Interventions: Drug: Elimite™ Cream (permethrin) 5%
- Test: Permethrin Cream, 5% (Experimental): Test: Permethrin Cream, 5% (Encube Ethicals)
  Interventions: Drug: Permethrin Cream, 5%

INTERVENTIONS:
Drug: Permethrin Cream, 5% — Permethrin Cream 5%
  Arms: Test: Permethrin Cream, 5%
Drug: Elimite™ Cream (permethrin) 5% — Permethrin Cream 5%
  Other Names: Elimite™ Cream
  Arms: Reference: Elimite™ Cream

SUMMARY:
Study to Evaluate the Therapeutic Equivalence of Permethrin Cream 5%in the Treatment of Scabies.

DETAILED DESCRIPTION:
A Randomized, Double-Blind, Parallel-Design, Multiple-Site Study to Evaluate the Therapeutic Equivalence of Permethrin Cream 5% (Encube Ethicals) Compared to Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.) in the Treatment of Scabies.

The objectives of this study are to:

1. Evaluate the therapeutic equivalence of the Test formulation, Permethrin Cream, 5% (Encube Ethicals) to the marketed product, Elimite™ Cream (permethrin) 5% (Prestium Pharma, Inc.) in patients with scabies.
2. Compare the safety of Test and Reference treatments in patients with scabies.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, 2 years of age or older.
2. If female and of childbearing potential, prepared to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., double barrier methods, intrauterine device (IUD), oral, transdermal or injected hormonal contraceptives). Female patients using hormonal contraceptives should have been on the same product/dosing regimen for at least 28 days before baseline and should not change this regimen during the study.
3. Signed informed consent that meets all criteria of current FDA and International Council for Harmonisation of Technical Requirements for Pharmaceuticals for Human Use (ICH) regulations. For patients who are considered minors in the state the study is being conducted (< 18 years in most states) the parent or legal guardian should sign the consent form and the child will be required to sign a patient "assent" form, as appropriate. Patients 11-17 years of age will read and sign an Independent Review Board (IRB)-approved assent form and patients 6-10 years of age will provide verbal assent. Patients 2-5 years of age will be exempt from providing assent based on the child's comprehension and cognitive skills.
4. Clinical diagnosis of active scabies by presence of a burrow and/or typical scabietic lesions at the classic sites of infestation.
5. Parasitological confirmation of clinical diagnosis with demonstration under light microscope of mites and/or their products (larvae, eggs or fecal material).
6. Symptom score of 2 or 3 on a 4-point rating scale of 0-3 for nocturnal itching/pruritus.
7. Ability to apply or have study product applied as directed. If patient is a child, then parent/guardian will apply study product to him/her.

Exclusion Criteria:

1. Patients who are pregnant, lactating, or planning to become pregnant during the study.
2. Any systemic or dermatologic disorder that, in the opinion of the Investigator, will interfere with the study results or increase the risk of adverse events (AEs).
3. Known hypersensitivity to permethrin cream or any of its components.
4. Use of any systemic or topical acaricide or ectoparasiticide within one month before Screening.
5. Patient has signs of a systemic infection or is receiving systemic therapy for an infectious disease.
6. Patients with severe cutaneous bacterial or fungal infections requiring therapy (including systemic and topical antibiotics) or coexisting dermatological disorder that could interfere with the diagnosis and subsequent monitoring of scabies) or heavily crusted with lesions consistent with Norwegian scabies.
7. Patients with an underlying immunodeficient state (including prolonged treatment with corticosteroids), immunosuppressive disorders requiring therapy, severe systemic disease and history of HIV infection.
8. Any condition, medical, psychological, or social, that, in the Investigator's opinion, would interfere with participation in the study.
9. Family members of employees of the clinic or Investigator.
10. Patients who, in the opinion of the Investigator, would be non-compliant with the requirements of the study protocol.
11. Patients whose close personal contacts will not or are not willing to comply with standard of care for Scabies management.
12. Receipt of any drug as part of a research study within 30 days before Screening.
13. History of seizures.
14. Use of systemic corticosteroids within two weeks before Screening.
15. Use of topical corticosteroids within one week before Screening.
16. Previous participation in this study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-11-11 (Actual); Study Completion 2017-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pratik Kamani, Study Director — Encube Ethicals Pvt. Ltd.
Locations (15):
- United States (10):
  - Applied Research Center of Arkansas, Little Rock, Arkansas
  - St. Josephs Clinical Research, Anaheim, California
  - Long Beach Clinical Trials, Long Beach, California
  - Havana Research Institute, Pasadena, California
  - Integrity Clinical Research Center, Inc., Hialeah, Florida
  - The Chappel Group Research, Kissimmee, Florida
  - Lenus Research & Medical Group, LLC, Sweetwater, Florida
  - DermDox Cetners for Dermatology, Hazleton, Pennsylvania
  - West Houston Clinical Research Services, Houston, Texas
  - Sun Research Instiute, San Antonio, Texas
- El Salvador (3):
  - Clinica Dermatologica/APF Research International, San Salvador
  - Clinica Dermatologica Y Cirugia de Piel/APF Research International, San Salvador
  - Clinica de la Doctora Laura Vargas, San Salvador
- Puerto Rico (2):
  - APF Research International, Aguas Buenas
  - APF Research International, Loíza

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Two hundred fifty-four (254) patients were randomized to study products. Thirteen (13) sites randomized patients into the study.The first patient was enrolled on 06/14/2017 and the last patient completed was on 10/30/2017. The time from first patient enrolled until last patient completed was approximately four months.
Pre-assignment Details: All eligible patients were randomized at visit 1 and received the study product with instructions for dosing at home.
Period: Overall Study
Arm/Group | Reference: Elimite™ Cream | Test: Permethrin Cream, 5%
Started | 129 | 125
Completed | 126 | 123
Not Completed | 3 | 2
Not completed — Withdrawal by Subject | 2 | 0
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Reference: Elimite™ Cream | Test: Permethrin Cream, 5% | Total
Number analyzed (Participants) | 129 | 125 | 254
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.7 (21.2) | 37.7 (22.4) | 39.2 (21.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 73 | 145
  Male | 57 | 52 | 109
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 96 | 97 | 193
  Not Hispanic or Latino | 33 | 28 | 61
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 14 | 15 | 29
  White | 109 | 108 | 217
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Puerto Rico | 6 | 6 | 12
  El Salvador | 63 | 62 | 125
  United States | 60 | 57 | 117
Baseline Severity Score of Nocturnal Itching Pretreatment [Count of Participants; unit: Participants]
  None | 0 | 0 | 0
  Mild | 0 | 0 | 0
  Moderate | 112 | 110 | 222
  Severe | 17 | 15 | 32
Baseline Severity of Lesion Count Infestation Pretreatment [Count of Participants; unit: Participants]
  Mild | 47 | 45 | 92
  Moderate | 68 | 57 | 125
  Severe | 14 | 23 | 37

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients in Each Treatment Group With Therapeutic Cure (Parasitological Cure Plus Clinical Cure) of Scabies
Description: Parasitological cure is defined as failure to demonstrate microscopically the presence of scabies infestation (i.e., no living mites, no viable mite eggs, and no mite fecal matter present).
  Clinical cure is defined as visual evidence of absence of new lesions and healing of original lesions, regardless the presence of post-scabietic nodules (i.e., post-scabietic nodules need not be considered as new lesions or persistence of old lesions).
Time Frame: Day 28 ± 4
Population: The Per Protocol (PP) population was used for the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference: Elimite™ Cream | Test: Permethrin Cream, 5%
Number analyzed (Participants) | 119 | 117
Participants | 83 | 86

2. Other Pre Specified Outcome: Number of Patients With a Therapeutic Cure That Completed Visit 2 Within 14 ± 2 Days and Visit 3 Within 28 ± 4 Days.
Description: as for outcome 1
Time Frame: Visit 2 Within 14 ± 2 Days and Visit 3 Within 28 ± 4 Days
Population: Patients who completed Visit 2 within 14 ± 2 days and Visit 3 within 28 ± 4 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reference: Elimite™ Cream | Test: Permethrin Cream, 5%
Number analyzed (Participants) | 110 | 110
Participants | 77 | 81

3. Other Pre Specified Outcome: Number of Patients With a Therapeutic Cure That Completed Visit 2 Within 14 ± 2 Days and Visit 3 Between Day 26 and Day 32, Inclusive.
Description: as for outcome 1
Time Frame: Visit 2 within 14 ± 2 days and Visit 3 between Day 26 and Day 32, inclusive.
Population: Number of patients with a Therapeutic Cure that completed Visit 2 within 14 ± 2 days and Visit 3 between Day 26 and Day 32, inclusive.
Measure: Count of Participants; unit: Participants
Arm/Group | Reference: Elimite™ Cream | Test: Permethrin Cream, 5%
Number analyzed (Participants) | 101 | 102
Participants | 68 | 75

4. Other Pre Specified Outcome: Number of Patients With a Therapeutic Cure That Completed Visit 2 Within 14 ± 2 Days and Visit 3 Within 28 ± 2 Days.
Description: as for outcome 1
Time Frame: Visit 2 Within 14 ± 2 Days and Visit 3 Within 28 ± 2 Days
Population: Patients who completed Visit 2 within 14 ± 2 days and Visit 3 within 28 ± 2 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reference: Elimite™ Cream | Test: Permethrin Cream, 5%
Number analyzed (Participants) | 95 | 100
Participants | 65 | 73

ADVERSE EVENTS:
Time Frame: 4.5 months
Arm/Group | Reference: Elimite™ Cream | Test: Permethrin Cream, 5%
All-Cause Mortality (participants affected / at risk) | 0/129 | 0/125
Serious Adverse Events (participants affected / at risk) | 0/129 | 1/125
Other Adverse Events (participants affected / at risk) | 7/129 | 7/125
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference: Elimite™ Cream (N=129) | Test: Permethrin Cream, 5% (N=125)
Left Foot Cellulitus (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Reference: Elimite™ Cream (N=129) | Test: Permethrin Cream, 5% (N=125)
Headache (Nervous system disorders) | 2 (2) | 2 (2)
Erythema In Helix Skin Of The Right Ear (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Pain In Extremity/Leg Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Enterocolitis/Acute Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Viral Upper Respiratory Tract Infection/Common Cold (Infections and infestations) | 0 (0) | 1 (1)
Bone Pain/Bone Ache (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Application Site Hypoaesthesia (General disorders) | 1 (1) | 0 (0) — Right Arm Numbness
Application Site Paraesthesia (General disorders) | 1 (1) | 0 (0) — Tingling Sensation In The Skin
Pharyngitis/Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
Application Site Rash/Rash (General disorders) | 1 (1) | 0 (0)
Abdominal Pain/Upper Epigastralgia (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the Clinical Trials Agreements between the sites and the Contract Research Organization, sites are instructed that the Investigator shall not publish, or seek to publish, either in whole or in part any results of the Study without the written consent.

DOCUMENTS (2):
  • Study Protocol (2017-11-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT03178942/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-02): https://cdn.clinicaltrials.gov/large-docs/42/NCT03178942/SAP_001.pdf